CLINICAL TRIAL: NCT01871701
Title: Clinical Trial to Investigate the Effect on Corrected QT Interval Prolongation by Psychotropic Drugs in Healthy Korean Adults After a Single Oral Administration of Escitalopram, Quetiapine, and Moxifloxacin
Brief Title: Clinical Trial to Investigate the Effect on Corrected QT Interval Prolongation by Psychotropic Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jae Yong Chung, Assistant Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CNSQT
Record Dates: First submitted 2012-12-05; First posted 2013-06-07 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: Corrected QT interval prolongation; Psychotropic drugs
MeSH Terms: interventions — Escitalopram; Tablets; Quetiapine Fumarate; Moxifloxacin; Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Quetiapine (Experimental): Quetiapine 100 mg (Seroquel, Tablet)
  Interventions: Drug: Quetiapine
- Moxifloxacin (Experimental): Moxifloxacin 400 mg (Avelox, Tablet)
  Interventions: Drug: Moxifloxacin
- Escitalopram (Experimental): Escitalopram 20 mg (Lexapro, Tablet)
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Water intake
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Escitalopram — Escitalopram
  Other Names: Escitalopram 20 mg (Lexapro, Tablet)
  Arms: Escitalopram
Drug: Quetiapine — Quetiapine
  Other Names: Quetiapine 100 mg (Seroquel, Tablet)
  Arms: Quetiapine
Drug: Moxifloxacin — Moxifloxacin
  Other Names: Moxifloxacin 400 mg (Avelox, Tablet)
  Arms: Moxifloxacin
Other: Placebo — Placebo
  Other Names: Water intake
  Arms: Placebo

SUMMARY:
To evaluate the corrected QT interval change(automatic-reading) after single oral administration of escitalopram, quetiapine and moxifloxacin versus placebo in healthy Korean Adults.

DETAILED DESCRIPTION:
Randomized, Open-label, Placebo-controlled, 4-way crossover study

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 20 - 40 years.
2. A body weight in the range of 50 kg (inclusive) - 90 kg (inclusive) and a body mass index (BMI) in the range 19.0 kg/m2 (inclusive) - 25.0 kg/m2 (inclusive).
3. Sufficient ability to understand the nature of the study and any hazards of participating in it. Provide written informed consent after being fully. informed about the study procedures.

Exclusion Criteria:

1. Presence or history of hypersensitivity or allergic reactions to drugs including investigational product (Escitalopram, Quetiapine, Moxifloxacin)) or other quinolone group antibiotics.
2. Subject judged not eligible for study participation by investigator.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Corrected QT interval prolongation | Predose (3 times) and 1, 2, 3, 4, 6, 8, 12, 16, 24 h, additional 26, 28, 32, 48 h after escitalopram dosing

SECONDARY OUTCOMES:
AUC (area under the plasma concentration-time curve) of escitalopram | Predose and 1, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48h postdose
  AUC, Cmax, Tmax, t1/2, CL/F
AUC (area under the plasma concentration-time curve)of quetiapine, moxifloxacin | Predose and 1, 2, 3, 4, 6, 8, 12, 16, 24 h postdose
  AUC, Cmax, Tmax, t1/2, CL/F

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Yong Chung, MD, PhD, Principal Investigator — Department of Clinical Pharmacology and Therapeutics, Seoul National University Bundang Hospital, Seongnam, Korea
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Gyounggi, South Korea